CLINICAL TRIAL: NCT04973501
Title: Evaluation of the Effect of the Physiotherapy on Mobility and Functional Disorders of the Musculoskeletal System in People With Multiple Sclerosis
Brief Title: Functional Disorders of the Musculoskeletal System in People With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Kamila Řasová, assoc. prof. Kamila Řasová, Ph.D., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EK-VP/25/0/2014/2
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Multiple Sclerosis; Rehabilitation; Musculoskeletal Complication
Keywords: Developmental kinesiology; Physiotherapy; Muscle imbalance; Musculoskeletal disorders
MeSH Terms: conditions — Multiple Sclerosis; Musculoskeletal Diseases | interventions — Methods

STUDY DESIGN:
Intervention Model Description: The study was designed as parallel group (outpatients) randomized comparison of two kinds of physiotherapeutic interventions.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual physiotherapeutic correction (MFK) Method (Experimental): The MFK was chosen for our clinical experience- it was developed in Czech Republic.The MFK Method consists of five established steps: anamnesis, assessment, diagnoses, treatment and checkup. In the course of all those steps, the computer MFK System software is used. This software allows us to display and visualize the patient´s functional muscle imbalance at the day of the assesment based on the assessment of muscle strength by manual muscle tests. Hereafter the physiotherapist performs muscle test and records results in the software. Then, the software visually describes the patient´s imbalance at the day of the assessment. Based on these diagnostic maps and the software suggestions the therapist chooses the body areas where the therapeutic techniques may be applied.
  Interventions: Behavioral: Manual physiotherapeutic correction (MFK) Method
- Dynamic Neuromuscular Stabilization (DNS) Method (Experimental): Dynamic Neuromuscular Stabilization (DNS) is a neurophysiological rehabilitative approach encompassing a set of functional tests assessing the quality of postural stabilization patterns and a treatment approach based on developmental kinesiology models. DNS diagnosis is based on comparison of the individual's postural stabilization pattern to the developmental stabilization pattern of healthy infants. The assessor uses DNS evaluation sheet to screen client's posture in 11 developmental positions if the patient can perform them all. If not, only the tests that the patient can perform sufficiently and safely serve for functional assessment. The strategy of DNS manual treatment is to utilize only those functional exercises in developmental positions that are the most suitable for the specific client. The goal is to improve spinal and joint stability by focusing on the global stabilization system consequently improving quality of movement and mobility.
  Interventions: Behavioral: Dynamic Neuromuscular Stabilization (DNS) Method

INTERVENTIONS:
Behavioral: Manual physiotherapeutic correction (MFK) Method — Patients undergo ambulatory physiotherapy :1-hour duration, twice a week for one month and once a week for next two months (16 therapies in total). Therapy was undertaken at the ambulatory section of the Department of Neurology, Kralovske Vinohrady University Hospital in Prague.
  Arms: Manual physiotherapeutic correction (MFK) Method
Behavioral: Dynamic Neuromuscular Stabilization (DNS) Method — Patients undergo ambulatory physiotherapy :1-hour duration, twice a week for one month and once a week for next two months (16 therapies in total).Therapy was undertaken at the Department of Rehabilitation and Sport Medicine, Motol University Hospital.
  Arms: Dynamic Neuromuscular Stabilization (DNS) Method

SUMMARY:
The randomized controlled trial is aimed to study the efficacy of treatment approaches based on developmental kinesiology models and its impact on balance, gait and mobility in people with mild to severe multiple sclerosis (pwMS). The main goal is to compare two out-patient physiotherapeutic methods, that will be attended 1-hour twice a week for one month and once a week for next two months (16 therapies in total). The efficacy will be assessed by a blinded independent clinical examiner using clinical examination and questionnaire survey one month before the therapy programme, immediately before and after the therapy and two months after termination of the therapy.

DETAILED DESCRIPTION:
The participants were randomly divided into two groups for three-month outpatient physiotherapeutic programme.

One group obtained treatment by MFK Method (Manual physiotherapeutic correction) and the second by DNS (Dynamic Neuromuscular Stabilization ). Both treatment methods were developed in the Czech Republic. All participants attended 1-hour MFK Method or DNS twice a week for one month and once a week for next two months (16 therapies in total).

The participants were examined three times - before the start of the physiotherapy program, immediately after its completion and six months apart.

ELIGIBILITY:
Inclusion Criteria:

* exact diagnosis of MS stated by neurologist
* Expanded Disability Status Scale (EDSS) ≥ 2 and ≤ 6,5
* no previous physiotherapy in six months
* no clinical relapses and changes in pharmacotherapy in the previous month or during the rehabilitation trial
* ability to undergo ambulatory physiotherapy

Exclusion Criteria:

* other neurological disease or conditions disabling movement (e.g. stroke, pregnancy, fracture)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) | six months
  The TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around, walk back to the chair, and sit down.
Berg Balance Scale (BBS) | six months
  14 items objective measure of static balance and risk of falls (0 the best, 56 the worse)
Dynamic Gait Index (DGI) | six months
  The DGI tests the ability of the participant to maintain walking balance while responding to different task demands, through various dynamic conditions.
  It includes eight items, walking on level surfaces, changing speeds, head turns in horizontal and vertical directions, walking and turning 180 degrees to stop, stepping over and around obstacles, and stair ascent and descent.
  Each item is scored on a scale of 0 to 3, with 3 indicating normal performance and 0 representing severe impairment.
  The best possible score on the DGI is a 24
Five times Sit to Stand test (5STS) | six months
  The test assesses time when people stand and sit repeatedly five times. The lower the time to complete the test the better the outcome of the test.
2-Minute Walk Test (2MWT) | six months
  The 2MWT is a simple measure of the distance a person can walk in two minutes. Rest breaks are allowed if needed. The person is encouraged to walk as fast as they can, safely, for two minutes. Walking aids can be used as needed e.g. for elderly people with a record made of walking aid used. If Assistive devices are used , they should be kept consistent and documented from test to test.
Symbol Digit Modalities Test (SDMT) | six months
  The SDMT involves a simple substitution task. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Because examinees can give either written or spoken responses, the test is well suited for use with individuals who have motor disabilities or speech disorders.
Four Square Step Test (FSST) | six months
  The subject is required to sequentially step over four canes set-up in a cross configuration on the ground.
  At the start of the test, the subject stands in Square 1 facing Square 2. The aim is to step as fast as possible into each square with both feet in the following sequence: Square 2, 3, 4, 1, 4, 3, 2, 1 (clockwise to counterclockwise) Test procedure may be demonstrated, one practice trial is allowed prior to administering the test.
  Two trials are then performed, and the better time (in seconds) is taken as the score.
  Timing starts when the first foot contacts the floor in Square 2 and finishes when the last foot comes back to touch the floor in Square 1.

SECONDARY OUTCOMES:
Questionnaires - The Fatigue scale for motor and cognitive functions (FSMC) | six months
  FSMC - is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue).
Questionnaires -Multiple Sclerosis Impact Scale (MSIS-29) | six months
  A 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on a day-to-day life in the past two weeks. All items have 5 response options: 1 "not at all" to 5" extremely". Each of the two scales is scored by summing the responses across items, then converting to a 0-100 scale where 100 indicates the greater impact of the disease on daily function (worse health).
Questionnaires - Euroqol-5 dimensions-5 levels health questionnaire | six months
  Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each of which has three severity levels that are described by statements appropriate to that dimension. A higher number means a worse quality of life.
Questionnaires -Multiple Sclerosis Walking Scale-12 (MSWS-12) | six months
  The Multiple Sclerosis Walking Scale is a self-assessment scale which measures the impact of MS on walking. It consists of 12 questions concerning the limitations to walking due to MS during the past 2 weeks. Each item can be answered with 5 options, with 1 meaning no limitation and 5 extreme limitation.
  A total score can be generated and transformed to a 0 to 100 scale by subtracting the minimum score possible (12) from the patient's score, dividing by the maximum score possible minus the minimum possible (60-12 or 48), and multiplying the result by 100.
Questionnaires - Rivermead Mobility (RMI) | six months
  The Rivermead Mobility Index is a measuring instrument for functional loss related to body mobility. It measures the patient's ability to move her or his own body.
  14-self-reported items
  1 direct observation item Items progress in difficulty Items are coded as either 0 or 1, depending on whether the patient can complete the task according to specific instructions Items receive a score of 0 for a "No" response and 1 for a "Yes" response Total scores are determined by summing the points for all items A maximum of 15 points is possible; higher scores indicate better mobility performance A score of "0" indicates an inability to perform any of the activities on the measure
Questionnaires- Activities-specific Balance Confidence Scale (ABC) | six months
  The patient is asked to rate their confidence in their balance, while performing 16 activities, on a percentage scale of 0 to 100, where 0 is a certainty of falling or becoming unstable and 100 is complete confidence in the patient's own ability to stay balanced.
  The final score is the average of the 16 individual scores for each activity.

CONTACTS AND LOCATIONS:
Overall Officials: Kamila Řasová, Ph.D., Principal Investigator — Charles University, Czech Republic